CLINICAL TRIAL: NCT03972514
Title: Prospective Observational Trial of the Impact of Radiation Dose on Brain Morphology, Volumetric Changes, Endocrine Function, and Neurocognitive Function Following Cranial Radiation Therapy in Children With Brain and Skull Base Tumors.
Brief Title: Observational Trial of the Impact of Radiation Dose in Children With Brain and Skull Base Tumors.
Status: Active, not recruiting | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Collaborators: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-LLB-HALL-001
Record Dates: First submitted 2019-04-25; First posted 2019-06-03 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor; Brain Cancer; Skull Base Tumor
Keywords: brain; pediatrics brain cancer; pediatrics; skull
MeSH Terms: conditions — Brain Neoplasms; Skull Base Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational clinical trial investigating the morphological and volumetric changes in the brain following cranial Radiation Therapy in pediatric patients with brain or skull base tumors.

DETAILED DESCRIPTION:
Brain injury is a known complication of cranial RT, but little is known about the factors that predispose patients to such injury. The brain is a highly interconnected organ linked through neuronal connections, cellular migration, and vascular supply and is endowed with exquisitely radiosensitive stem cell niches responsible for neuro-regeneration. To date, the effects of brain radiation have been quantified in few brain substructures. The majority of publications on this topic have focused on regions receiving higher doses. Even low dose radiation exposure, however has global implications on brain development and function, and its effects are less well studied. It is increasingly recognized that radiation damage to one brain region can potentially affect brain development more broadly. This has important implications on RT planning and the potential for understanding its long-term effects.

In this protocol, the investigators aim to measure serum inflammatory cytokine levels and other molecular biomarkers at baseline and post-exposure in an exploratory manner to investigate potential associations with the risk of developing volumetric changes in the brain and radiation-induced toxicities.

This study will observe sixty (60) patients under the age of 21 with brain or base of skull tumor. The study team will observe the effect of radiation therapy per the study protocol versus standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient (parent) must give study-specific informed consent on an IRB-approved consent prior to any research related procedures or study treatment. Written assent will be obtained as per Institutional guidelines.
* Patients (Age equal to or less than 35 years old) that are planned to receive photon or proton RT to the brain according to standard of care are eligible to participate.
* Patients that are planned to receive fractionated RT at 1.2-2.0 Gy RBE dose per fraction per standard of care are eligible to participate. If patients are planned to receive an alternative dose/fractionation regimen, then they should be treated according to standard of care and should not be enrolled.
* Zubrod/Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1

Exclusion Criteria:

* Patient cannot undergo MRI without contrast as per standard of care
* Patient and family do not speak English or Spanish
* Patient receiving treatment with non-curative intent
* Patients with an expected 3-year overall survival less than 50%

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study sample size will be 60 patients. This sample size was selected to ensure an adequate distribution of primary tumor diagnoses and dosimetric variation in major brain substructures treated based on tumor location/brain regions treated. The estimated case distribution based on historical data from 2007-2015 will be: Craniopharyngioma 20%, Ependymoma 20%, Low Grade Glioma 20%, Medulloblastoma/PNET 15%, Sarcoma 10%, Other 15%.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Measure temporal changes in brain volumes | Baseline, 6 Months, 12 months, 18 months, 24 months and 3-5 years
  Measure temporal changes in brain volumes after exposure to therapeutic RT and to correlate these changes with absorbed dose.
Measure temporal changes in morphometry | Baseline, 6 Months, 12 months, 18 months, 24 months and 3-5 years
  Measure temporal changes in morphometry after exposure to therapeutic RT and to correlate these changes with absorbed dose.

SECONDARY OUTCOMES:
Morphometric changes in the brain | Baseline, 6 Months, 12 months, 18 months, 24 months and 3-5 years
  The secondary aims for this study are to correlate morphometric changes in the brain with the development of late treatment-related effects, including measurable neurocognitive, endocrine, and quality of life effects.

OTHER OUTCOMES:
Measure molecular biomarkers | Baseline, 6 Months, 12 months, 18 months, 24 months and 3-5 years
  Serum pro-inflammatory and anti-inflammatory cytokine levels will be measured at baseline and during follow-up as part of an exploratory hypothesis-generating correlate study to analyze potential associations with risk of radiation-induced toxicities and volumetric changes in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Hall, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Miami Cancer Institute Website — https://baptisthealth.net/cancer-care/home